CLINICAL TRIAL: NCT07223632
Title: The Treatment of Charcot-Marie-Tooth Disease, Axonal, Type 2S (CMT2S) in an Individual Patient With Confirmed IGHMBP2 Intronic Cryptic Splice Variant C. 1235+894C>A That is Amenable to Antisense Oligonucleotide (ASO)-Mediated Correction of IGHMBP2 Splicing
Brief Title: Treatment of Charcot-Marie-Tooth Disease, Axonal, Type 2S (CMT2S) in an Individual Patient
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP-VCA-894A-2101
Record Dates: First submitted 2025-10-27; First posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Charcot Marie Tooth Disease (CMT); Neuromuscular Diseases (NMD)
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Neuromuscular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VCA-894A (Experimental)
  Interventions: Drug: VCA-894A

INTERVENTIONS:
Drug: VCA-894A — intrathecal antisense oligonucleotide injection

SUMMARY:
This is an 'N of 1', open-label, single center study to evaluate the safety of therapy with VCA-894A, an ASO designed to rescue and restore the activity of IGHMBP2, when administered by intrathecal injection.

ELIGIBILITY:
Inclusion Criteria:

* Ability and acceptance to provide written informed consent.
* Genetically confirmed diagnosis of CMT2S with confirmed IGHMBP2 intronic cryptic splice variant c. 1235+894C>A.

Exclusion Criteria:

* Significant clinical deterioration of the patient's neurologic status, as judged by the Investigator.
* Non-reversible conditions that are contraindications to lumbar puncture.
* Pregnancy, recent pregnancy (within 6 weeks), or women who are breastfeeding.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of safety of therapy with VCA-894A when administered via intrathecal injection, as measured by the incidence of adverse events. | 295 days
  Safety will be assessed by determining the incidence, severity, and dose relationship of adverse events that are related to treatment with VCA-894A.
Assessment of CMT2S symptoms following chronic administration of intrathecal VCA-894A, as determined by the change in the Revised Upper Limb Module for Spinal Muscular Atrophy (RULM). | 295 days
  The Revised Upper Limb Module for Spinal Muscular Atrophy (RULM) scores range from a minimum of 0 to a maximum of 37 points, with higher scores indicating better upper limb function.
Assessment of CMT2S symptoms following chronic administration of intrathecal VCA-894A, as determined by the change in the Hammersmith Functional Motor Scale - Expanded (HFMSE). | 295 days
  The Hammersmith Functional Motor Scale - Expanded (HFMSE) scores range from a minimum of 0 to a maximum of 66 points, with higher scores indicating greater motor functioning.

SECONDARY OUTCOMES:
Rescue of IGHMBP2, as determined by the change in IGHMBP2 mRNA expression from baseline. | 295 days
  IGHMBP2 mRNA, which is the target of VCA-894A therapy, will be measured in both the cerebrospinal fluid (CSF) and blood by qPCR relative expression.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanda Investigational Site, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smieszek S, Przychodzen B, Tyner C, Johnson C, Bai H, Kwon JM, Hagan DW, Niccum C, Brighton R, Hawkins K, Aiken R, Nawaz A, Guo X, Hickman J, Polymeropoulos CM, Birznieks G, Polymeropoulos MH. Potential ASO-based personalized treatment for Charcot-Marie-Tooth disease type 2S. Mol Ther Nucleic Acids. 2025 Feb 4;36(1):102479. doi: 10.1016/j.omtn.2025.102479. eCollection 2025 Mar 11. PMID 40060931